CLINICAL TRIAL: NCT01987219
Title: The Effects of Bronchodilator Therapy On Respiratory and Autonomic Function in Patients With Familial Dysautonomia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13-00004
Record Dates: First submitted 2013-11-05; First posted 2013-11-19 (Estimated); Results first posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-04

CONDITIONS: Familial Dysautonomia
Keywords: familial dysautonomia
MeSH Terms: conditions — Dysautonomia, Familial | interventions — Albuterol; Ipratropium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Albuterol-sulphate (Active Comparator): Albuterol-sulphate (Proventil ®) Beta-2-adrenergic agonist 2.5 mg 3 cc inhalation Peak effect 15 - 30 mins. Mean duration of effect 3 hours
  Interventions: Drug: Albuterol-sulphate
- Ipratropium-bromide (Atrovent ®) (Active Comparator): IpratroAnti-cholinergic(Atrovent ®) 500 mcg 3 cc inhalation Peak effect 30 - 90 mins. Duration of effect 2 - 4 hours.pium-bromide
  Interventions: Drug: Ipratropium-bromide
- Placebo (Placebo Comparator): Placebo Saline solution 3 cc NA
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Albuterol-sulphate — Beta-2-adrenergic agonist 2.5 mg 3 cc inhalation Peak effect 15 - 30 mins. Mean duration of effect 3 hours
  Other Names: (Proventil ®)
  Arms: Albuterol-sulphate
Drug: Ipratropium-bromide — Anti-cholinergic 500 mcg 3 cc inhalation Peak effect 30 - 90 mins. Duration of effect 2 - 4 hours.
  Other Names: (Atrovent ®)
  Arms: Ipratropium-bromide (Atrovent ®)
Other: placebo — Saline solution 3 cc NA
  Arms: Placebo

SUMMARY:
Evaluate the effects of bronchodilator therapy on respiratory function. Our overall goal is to determine whether, in patients with familial dysautonomia (FD), there is a component of airway obstruction that is reversible. To this end, we will evaluate airway resistance before and after receiving the anti-cholinergic ipratropium (Atrovent ®) and the beta-2-agonist albuterol (ProVentil®/Ventolin®). We predict that the response to either drug will depend on the underlying level of sympathetic and parasympathetic activity and airway tone. We will then determine the cardiovascular effects of inhaled ipratropium and albuterol in patients with FD. Because patients with FD have fewer sympathetic neurons and denervation supersenstivity, we predict that following albuterol inhalation, there will be non-selective activation of alpha-1-adrenergic receptors. Furthermore, because of a congenital defect in the afferent baroreceptor neurons that sense blood pressure, we suspect that the resulting vasoconstriction will be unopposed leading to a pressor effect. We hypothesize that inhalation of the anti-cholinergic ipratopium will produce little rise in heart rate, due to the extent of parasympathetic denervation to the heart.

DETAILED DESCRIPTION:
Familial dysautonomia (FD) is a rare fatal autosomal recessive disease caused by a deficiency of the protein IKAP.1 This results in a selective developmental defect that affects mostly afferent (sensory) neurons including those in the dorsal root ganglia and cranial nerves.2, 3 We have shown recently that the protein deficiency impairs the development of afferent baroreceptor pathways, leaving the sympathetic efferent neurons reduced in number but functionally active. This results in the complete failure to detect and buffer fluctuations in blood pressure leading to volatile hypertension. In addition to the afferent baroreflex pathways, the deficiency of IKAP during embroyogenesis also affects the function of the chemoreflex pathways. As a result, patients fail to increase ventilation adequately in response to hypoxia and hypercapnia.4 As well as the impairment of the neurological mechanisms that regulate breathing, patients with FD also have a combination of obstructive, restrictive and probably also neuromuscular lung disease. Failure to coordinate swallowing results in recurrent bouts of aspiration pneumonia occurring from birth.5, 6 Imaging studies show that almost all patients with FD have bronchial wall thickening, atelectasis and almost 30% have bronchiectasis7. Pulmonary function tests show air flow limitation and associated lung restriction with reduction in diffusion capacity12. Sudden attacks of asthma like wheezing are common 8 and frequently associated with emotional upset,5 a time when sympathetic outflow to the vasculature is increased heightened.3 There is also a component of restrictive lung disease, with a very high incidence of scoliosis, which frequently begins at an early age. Complicating matters further, many patients opt to undergo spine fusion surgery, 9 which could potentially worsen further chest wall compliance.10 Patients with FD also lack muscle spindles, 2 making it likely that they have neuromuscular abnormalities arising from the absence of proprioceptive feedback from the respiratory muscles involved in the coordination of breathing.

Severe respiratory disease is a leading cause of death in patients with FD and many are treated empirically with inhaled bronchodilators. It is not known, however, whether these drugs are effective at reversing increased airway resistance. Hence, there is an urgent need to understand if the short acting beta-2-adrenergic agonist albuterol and the anticholinergic ipratropium, are effective bronchodilators. Furthermore, because treatment with these agents has potential cardiovascular side effects, we will also analyze their effects on blood pressure, heart rate and cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of familial dysautonomia (Riley-Day syndrome, hereditary sensory and autonomic neuropathy type III) 2. Ages 12 and older: Bronchodilators are routinely used in young children with FD therefore they should be included in this study. The spirometry maneuver is highly dependent on patient cooperation and effort, and FD patients already have limitations that make the spirometry maneuver more problematic to perform such as difficulty with mouth closure and drooling. Therefore, we believe age 12 is a suitable age for FD patients to be included in this study, though in the general population reliable results can be obtained from the age of 6 and sometimes even younger.

  3. Patients using Albuterol or Ipratroprium will be included in the study but will be instructed not to take the 24 hours prior to the testing. It is a common practice in clinical medicine to withhold the inhalation drugs prior to performing pulmonary function tests in order to evaluate the response to bronchodilators, an integral part of the test. Patients with an acute respiratory exacerbation will not be enrolled, as withholding bronchodilators would not be advisable.

  4. Patients who are taking medications that might affect autonomic function such as anti-hypertensives, beta-blockers, midodrine and florinef will be included in the study and we will record current medication regimen and the time the medication was taken.

Exclusion Criteria:

- 1. Patients who last used inhaled anti-cholinergics or beta-2-agonists within 4-half lives of the drug.

2. Patients with an acute respiratory illness 3. Patients who have had lobectomies. 4. Patients using oxygen therapy throughout the day. 5. Patients who are unable to comply with the study requirements.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifteen patients with Familial Dysautonomia were enrolled into the study between March 2013 and December 2015. The study was conducted at the NYU Dsyautonomia Center and Israeli FD center.
Groups:
- Ipratropium; Alubterol; Placebo: Participants in this group received ipratropium followed by albuterol followed by placebo
- Albuterol; Placebo; Ipratropium: Participants in this group received albuterol followed by placebo followed by ipratropium
- Albuterol; Ipratropium; Placebo: Participants in this group received albuterol followed by ipratropium followed by placebo
- Placebo; Ipratropium; Albuterol: Participants in this group received placebo followed by ipratropium followed by albuterol
- Placebo; Albuterol; Ipratropium: Participants in this group received placebo followed by albuterol followed by ipratropium
- Ipratropium; Placebo; Albuterol: Participants in this group received ipratropium followed by placebo followed by albuterol
Period: Overall Study
Arm/Group | Ipratropium; Alubterol; Placebo | Albuterol; Placebo; Ipratropium | Albuterol; Ipratropium; Placebo | Placebo; Ipratropium; Albuterol | Placebo; Albuterol; Ipratropium | Ipratropium; Placebo; Albuterol
Started | 2 | 2 | 7 | 2 | 1 | 1
Completed | 2 | 2 | 6 | 2 | 1 | 1
Not Completed | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipratropium; Alubterol; Placebo | Albuterol; Placebo; Ipratropium | Albuterol; Ipratropium; Placebo | Placebo; Ipratropium; Albuterol | Placebo; Albuterol; Ipratropium | Ipratropium; Placebo; Albuterol | Total
Number analyzed (Participants) | 2 | 2 | 7 | 2 | 1 | 1 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Between 18 and 65 years | 2 | 2 | 5 | 2 | 1 | 1 | 13
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 0 | 0 | 0 | 7
  Male | 0 | 1 | 3 | 2 | 1 | 1 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  White, not of Hispanic-American Origin | 2 | 2 | 7 | 2 | 1 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Forced Vital Capacity
Description: FVC is a measure of the amount of air exhaled, and is measured in liters of air per second. The percentage in the change in the amount of air exhaled from baseline, measured in liters of air per second. Increase in the percentage of air exhaled from baseline indicates improvement in respiratory function.
Time Frame: Pre and 30 minutes post study drug administration
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Albuterol-sulphate | Ipratropium-bromide (Atrovent ®) | Placebo
Number analyzed (Participants) | 15 | 15 | 14
percentage change from baseline | 5.5 (13.6) | 4.7 (10.9) | 0.9 (10.7)

2. Primary Outcome: Change in Respiratory Function (Airway Resistance at 5 Hz) From Baseline
Description: The percentage change in respiratory function from baseline is measured in percentage change in Resistance, kPa/(L/s).
Time Frame: Pre and 30 minutes post study drug administration
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Albuterol-sulphate | Ipratropium-bromide (Atrovent ®) | Placebo
Number analyzed (Participants) | 15 | 15 | 14
percentage change from baseline | -22.7 (18.6) | -19.5 (15.5) | -1.1 (12.5)

3. Secondary Outcome: Change in Forced Expiratory Volume (FEV) From Baseline
Description: Forced expiratory volume is measured in liters of air per second. FEV was measured during the first second of exhalation.
Time Frame: Pre and 30 post study drug admistration
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Albuterol-sulphate | Ipratropium-bromide (Atrovent ®) | Placebo
Number analyzed (Participants) | 15 | 15 | 14
percentage change from baseline | 7.69 (12.06) | 4.81 (9.9) | -0.9 (7.6)

4. Secondary Outcome: Change in Forced Expiratory Flow Between 25-75% (FEF25-75)
Description: FEF25-75 is measured in liters of air per second at 25-75%
Time Frame: pre and 30 minutes post intervention
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Albuterol-sulphate | Ipratropium-bromide (Atrovent ®) | Placebo
Number analyzed (Participants) | 15 | 15 | 14
percentage change from baseline | 14.7 (30.6) | 11.5 (36.1) | -2.99 (23.3)

ADVERSE EVENTS:
Description: Serious and Other [Not Including Serious] Adverse Events were not collected/assessed.
Arm/Group | Albuterol-sulphate | Ipratropium-bromide (Atrovent ®) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes